CLINICAL TRIAL: NCT02349087
Title: Integrating EEG Into Acute Medicine: EEG in Resuscitated In-hospital Patients
Brief Title: EEG in Resuscitated In-hospital Patients
Status: Terminated | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KUH507T010
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Sudden Cardiac Arrest; Seizures
Keywords: EEG; cardiac arrest; resuscitation; seizures
MeSH Terms: conditions — Death, Sudden, Cardiac; Seizures; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Acute EEG with fast applicable EEG electrode

SUMMARY:
In Kuopio University Hospital Department of Clinical Neurophysiology there have been designed a fast EEG electrode, that is suitable for acute emergency use. This study will address the clinical use of acute EEG with this fast EEG electrode in in- hospital patients who have been resuscitated due to cardiac arest. After resuscitation patients will be treated in ICU and EEG will be recorded for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Resuscitated in-hospital patients

Exclusion Criteria:

* Patients with Do Not Attempt to Resuscitate-decision
* Patients who are not going to be treated in ICU after resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- hospital resuscitated patients, who are going to be treated in ICU after ROSC. Patients with Do Not Attempt to Resuscitate -decision will not be included.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
24 hours of EEG monitoring starting from resuscitation and quantity of non-convulsive status epilepticus found | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Esa Mervaala, MD, PhD,prof, Study Director — Clinical Neurophysiology
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland